CLINICAL TRIAL: NCT01418118
Title: An Assessment of the Effects of Pressors on Graft Blood Flow After Free Tissue Transfer Surgery: A Randomised Study
Brief Title: Assessment of the Effects of Pressors on Graft Blood Flow After Free Tissue Transfer Surgery
Acronym: Free4Flow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Mr SR Watt-Smith, Oxford Radcliffe Hospitals NHS Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-000073-37 5579; 2008 000073 37 (EudraCT Number); 08/H0606/31 (Other: Oxfordshire Research Ethics Committee)
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Oral Cancer; Head and Neck Cancer; Free Flap; Hypotension
Keywords: noradrenaline; norepinephrine; epinephrine; adrenaline; dobutamine; dopexamine; inotrope; pressor; sympathomimetic; free flap; transplantation; free tissue transfer; microsurgery; survival
MeSH Terms: conditions — Mouth Neoplasms; Head and Neck Neoplasms; Hypotension | interventions — Epinephrine; Norepinephrine; Dobutamine; dopexamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pressors (Experimental): Epinephrine, Norepinephrine, Dobutamine, Dopexamine
  Interventions: Drug: Epinephrine; Drug: Norepinephrine; Drug: Dobutamine; Drug: Dopexamine

INTERVENTIONS:
Drug: Epinephrine — 0.2mcg/kg/min maximum infusion; to increase mean arterial pressure by 30mmHg
Drug: Norepinephrine — Maximum infusion of 0.2mcg/kg/min, to increase mean arterial pressure by 30mmHg
Drug: Dobutamine — Maximum infusion rate of 8mcg/kg/min to increase mean arterial pressure by 30mmHg
Drug: Dopexamine — Maximum infusion rate of 5mcg/kg/min to increase mean arterial pressure by 30mmHg

SUMMARY:
Following surgery to remove tumours of the head and neck, patients undergo reconstruction with free flaps - tissue that is taken from elsewhere in the body and given a new blood supply by attaching it to vessels in the neck. Following this type of surgery, patients often need medication to maintain their blood pressure in the intensive care unit. The effect of these drugs on the transplanted tissues is unknown. This study investigates the effects of four commonly used drugs on free flap perfusion.

DETAILED DESCRIPTION:
The optimal sympathomimetic drug to support blood pressure without adverse vasoconstriction of free flap circulation remains unknown. This study examined the effects of four agents (epinephrine, norepinephrine, dobutamine and dopexamine) on free flaps following resection of head and neck cancer.

Twenty five patients were recruited to the study. Each patient received an infusion of the four drugs in a random order with an intervening washout period between drugs, at four infusion rates. Continuous free flap skin blood flow monitoring was performed using laser Doppler velocimetry, with a second sensor on normal skin acting as a control. Global cardiovascular variables were monitored using the LiDCO Rapid pulse contour analysis system.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing free tissue transfer surgery at the John Radcliffe Hospital wih planned post-operative admission to the intensive care unit.

Exclusion Criteria:

* Pregnancy
* Weight >100kg
* Contraindications to pressor infusions
* Overnight ventilation not indicated

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Absolute change in transfer function (flap vascular resistance) after pressor infusion. | Post infusion (at 4 hours)

SECONDARY OUTCOMES:
Relative change in transfer function after pressor infusion compared with "normal" tissue. | Post infusion (at 4 hours)
Change in flap flow after pressor infusion | Post infusion (at 4 hours)
Differences in frequency spectrum of skin blood flow between flaps and "normal" tissue before and after pressor infusion. | Post infusion (at 4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Watt-Smith, FDSRCS, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Eley KA, Young JD, Watt-Smith SR. Epinephrine, norepinephrine, dobutamine, and dopexamine effects on free flap skin blood flow. Plast Reconstr Surg. 2012 Sep;130(3):564-570. doi: 10.1097/PRS.0b013e31825dbf73. PMID 22929242